CLINICAL TRIAL: NCT00266266
Title: Human Papilloma Virus DNA Self-Test
Acronym: HPV
Status: Completed | Type: Observational
Sponsor: University of Louisville (Other)
Collaborators: James Graham Brown Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 529.03
Record Dates: First submitted 2005-12-15; First posted 2005-12-16 (Estimated); Last update posted 2017-12-29 (Actual); Status verified 2017-12

CONDITIONS: Papilloma Virus, Human
Keywords: Human Papilloma Virus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
HPV DNA testing by a clinician has been shown to be highly sensitive in detecting cervical disease. Can we prove that HPV self-testing will be sufficiently sensitive to detect disease in high risk population who for various reasons would not have routine pap smear screening?

DETAILED DESCRIPTION:
Women between the ages of 18 years to post-menopausal with documented abnormal pap smear atypical squamous cells of undetermined significance and higher will be enrolled into the study. Patients will be taught how to collect vaginal samples with dacron swab and vaginal tampons by means of instructional video and manufacturer's instruction guide respectively. Physicians will perform pap smear and colposcopy. All samples will be sent to the University of Louisville lab for processing for HPV DNA detection by Hybrid capture 2 method.

ELIGIBILITY:
Inclusion Criteria:

Abnormal pap smear ASCUS or higher

Age 18-postmenopausal

Exclusion Criteria:

Less than 18 years old

Prior hysterectomy

Pregnancy

Use of corticosteroids

HIV positive

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Abnormal pap smear ASCUS or higher
  Age 18-postmenopausal
Sampling Method: Probability Sample
Enrollment: 171 (Actual)
Dates: Start 2004-01; Primary Completion 2008-10 (Actual); Study Completion 2008-10 (Actual)

PRIMARY OUTCOMES:
HPV DNA self-testing device to detect disease in patients with abnormal Pap smear | Patient will self-test immediately prior to their standard physician papsmear
  To assess the concordance of HPV DNA self-testing device to detect disease in patients with abnormal Pap smear. Patients with a positive HPV Self-test by vaginal swab or vaginal tampon will be compared to the physician test results for concordance. Following patient self-sample collection, physician will collect cervical samples using a spatula. A self testing device which patients can use at their convenience will be beneficial in decreasing the incidence of cervical cancer in Kentucky.

CONTACTS AND LOCATIONS:
Overall Officials: Robert Edwards, MD, Principal Investigator — University of Louisville,James Graham Brown Cancer Center
Locations (1):
- James Graham Brown Cancer Center, Louisville, Kentucky, United States